CLINICAL TRIAL: NCT03305016
Title: fliGHt: A Multicenter, Phase 3, Open-Label, 26-Week Trial Investigating the Safety, Tolerability and Efficacy of TransCon hGH Administered Once Weekly in Children With GHD
Brief Title: A Safety, Tolerability and Efficacy Study of TransCon hGH in Children With Growth Hormone Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ascendis Pharma Endocrinology Division A/S (Industry)
Responsible Party: Sponsor
Organization: Ascendis Pharma A/S (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TransCon hGH CT-302; U1111-1199-8218 (Other: WHO UTN)
Record Dates: First submitted 2017-10-04; First posted 2017-10-09 (Actual); Results first posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Growth Hormone Deficiency, Pediatric; Endocrine System Diseases; Hormone Deficiency; Pituitary Diseases
Keywords: Human Growth Hormone; hGH; GHD; rhGH; Pediatric Growth Hormone Deficiency; Long Acting Growth Hormone; Somatropin; Prodrug; Growth Failure; Growth Hormone Replacement Therapy; Sustained Release Growth Hormone; Growth Hormone Deficiency; TransCon GH
MeSH Terms: conditions — Dwarfism, Pituitary; Endocrine System Diseases; Pituitary Diseases; Failure to Thrive

STUDY DESIGN:
Intervention Model Description: All study participants will receive TransCon hGH
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TransCon hGH (Experimental): Once weekly subcutaneous injection of TransCon hGH
  Interventions: Drug: TransCon hGH

INTERVENTIONS:
Drug: TransCon hGH — Once weekly subcutaneous injection at a starting dose of 0.24 mg/kg/week

SUMMARY:
A 26 week trial of TransCon hGH, a long-acting growth hormone product, administered once-a-week. Approximately 150 children (males and females) with growth hormone deficiency (GHD) will be included. All study participants will receive TransCon hGH. This is a global trial that will be conducted in, but not limited to, the United States, Canada, Australia, and New Zealand.

ELIGIBILITY:
Inclusion Criteria:

1. Investigator-determined GHD diagnosis prior to the historical initiation of daily hGH therapy.
2. 6 months to 17 years old, inclusive, at Visit 1

   1. If 3 to 17 years old, are taking daily hGH at a dose of ≥ 0.20 mg hGH/kg/week for at least 13 weeks but no more than 130 weeks prior to Visit 1
   2. If ≥ 6 months but < 3 years old, are either hGH treatment-naïve or are taking daily hGH at a dose of ≥ 0.20mg hGH/kg/week for no more than 130 weeks prior to Visit 1
3. Tanner stage < 5 at Visit 1
4. Open epiphyses (bone age ≤14.0 years for females or ≤16.0 years for males)
5. Written, signed, informed consent of the parent or legal guardian of the subject and written assent of the subject as required by the IRB/HREC/IEC

Exclusion Criteria:

1. Weight of < 5.5 kg or > 80 kg at Visit 1
2. Females of child-bearing potential
3. History of malignant disease
4. Any clinically significant abnormality likely to affect growth or the ability to evaluate growth (eg, chronic diseases or conditions such as renal insufficiency, spinal cord irradiation, hypothyroidism, active celiac disease, malnutrition or psychosocial dwarfism)
5. Poorly-controlled diabetes mellitus (HbA1c >8.0%) or diabetic complications
6. Known neutralizing antibodies against hGH
7. Major medical conditions, unless approved by Medical Monitor
8. Pregnancy
9. Presence of contraindications to hGH treatment
10. Likely to be non-compliant with respect to trial conduct (in regards to the subject and/or the parent/legal guardian/caregiver)
11. Participation in any other trial of an investigational agent within 30 days prior to Visit 1
12. Prior exposure to investigational hGH

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 146 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee D Shu, MD, Study Director — Ascendis Pharma, Inc.; David B Karpf, MD, Study Director — Ascendis Pharma, Inc.
Locations (24):
- United States (21):
  - University of Alabama, Birmingham, Alabama
  - Neufeld Medical Group Inc., Los Angeles, California
  - Center of Excellence in Diabetes and Endocrinology, Sacramento, California
  - Rocky Mountain Pediatric Endocrinology, Centennial, Colorado
  - Nemours Children's Health System, Jacksonville, Florida
  - Orlando Health Inc., Orlando, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - University of Iowa, Iowa City, Iowa
  - Children's Minnesota, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - NYU Winthrop Hospital, Mineola, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Diabetes and Endocrine Center, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Children's Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - University of Virginia Children's Hospital, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
- Monash Children's Hospital, Clayton, Victoria, Australia
- Stollery Children's Hospital, Edmonton, Alberta, Canada
- The Liggins Institute, The University of Auckland, Grafton, Auckland, New Zealand

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 162 subjects were screened for entry into this trial; of these, 16 subjects did not meet eligibility criteria and were considered screen failures.
Groups:
- Lonapegsomatropin: Once weekly subcutaneous injection of lonapegsomatropin (TransCon hGH) at a starting dose of 0.24 mg/kg/week
Period: Overall Study
Arm/Group | Lonapegsomatropin
Started | 146
Completed | 144
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Lonapegsomatropin
Number analyzed (Participants) | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.6 (3.9)
Age, Customized [Count of Participants; unit: Participants]
  Age, Categorical:: <3 years | 4
  Age, Categorical:: ≥3 and <6 years | 20
  Age, Categorical:: ≥6 to <11 years (girls) or ≥6 to <12 years (boys) | 55
  Age, Categorical:: ≥11 years (girls) or ≥12 years (boys) | 67
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 110
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 124
  Unknown or Not Reported | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 6
  Race: Black or African American | 3
  Race: Native Hawaiian or Other Pacific Islander | 2
  Race: White | 124
  Race: More than one race | 2
  Race: Unknown | 9
Height [Mean (Standard Deviation); unit: cm] | 132.4 (22.5)
Height SDS [Mean (Standard Deviation); unit: standard deviation score] — Height Standard Deviation Score (SDS) is the number of standard deviations above or below the mean height for age and sex. Height SDS was derived using the LMS method as ((Height/M)^L)-1)/(L x S), where M = median, S = generalized coefficient of variation, and L = power in the Box-Cox transformation, the M, S, L values were obtained from 2000 CDC growth charts for the United States. A Standard Deviation Score of 0 represents the population mean.
  standard deviation score | -1.42 (0.84)
Weight [Mean (Standard Deviation); unit: kg] | 32.3 (14.2)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 17.5 (3.0)
IGF-1 SDS [Mean (Standard Deviation); unit: standard deviation score] — IGF-1 Standard Deviation Score (SDS) is the number of standard deviations above or below the mean Insulin-like Growth Factor 1 (IGF-1) level for age and sex. IGF-1 SDS was derived using the LMS method as ((IGF-1/M)^L)-1)/(L x S), where M = median, S = generalized coefficient of variation, and L = power in the Box-Cox transformation, the M, S, L values were obtained from Bidlingmaier et al. (2014). A Standard Deviation Score of 0 represents the population mean.
  standard deviation score | 0.85 (1.29)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events [Safety and Tolerability]
Description: Safety and tolerability of weekly lonapegsomatropin (TransCon hGH) treatment
Time Frame: 26 weeks
Population: The Full Analysis Set included all subjects who received at least 1 dose of trial drug during the trial and who had any follow-up data.
Measure: Count of Participants; unit: Participants
Arm/Group | Lonapegsomatropin
Number analyzed (Participants) | 146
Participants
  TEAE | 83
  Related TEAE | 6
  Serious TEAE | 1
  Related Serious TEAE | 0

2. Secondary Outcome: Annualized Height Velocity (AHV) at 26 Weeks of Weekly Lonapegsomatropin Treatment
Description: Annualized height velocity (AHV) at 26 weeks of weekly lonapegsomatropin (TransCon hGH) treatment. The AHV at each visit was modeled using ANCOVA adjusting for baseline age, peak GH levels (log transformed) at diagnosis, delta average-parental height SDS, prior GH dose level (log transformed), and prior GH dose duration (log transformed) as covariates and gender as a factor. Subjects who did not take prior GH treatment were not included in the model.
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: cm/year
Arm/Group | Lonapegsomatropin
Number analyzed (Participants) | 144
cm/year | 8.72 (0.24)

3. Secondary Outcome: Number of Subjects With IGF-1 Standard Deviation Score (SDS) in the Range of 0.0 to +2.0 at 26 Weeks of Weekly Lonapegsomatropin Treatment
Description: IGF-1 Standard Deviation Score (SDS) is the number of standard deviations above or below the mean Insulin-like Growth Factor 1 (IGF-1) level for age and sex. IGF-1 SDS was derived using the LMS method as ((IGF-1/M)^L)-1)/(L x S), where M = median, S = generalized coefficient of variation, and L = power in the Box-Cox transformation, the M, S, L values were obtained from Bidlingmaier et al. (2014). A Standard Deviation Score of 0 represents the population mean.
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lonapegsomatropin
Number analyzed (Participants) | 142
Participants | 74

4. Secondary Outcome: Change in Height Standard Deviation Scores (SDS) at 26 Weeks of Weekly Lonapegsomatropin Treatment
Description: Height Standard Deviation Score (SDS) is the number of standard deviations above or below the mean height for age and sex. Height SDS was derived using the LMS method as ((Height/M)^L)-1)/(L x S), where M = median, S = generalized coefficient of variation, and L = power in the Box-Cox transformation, the M, S, L values were obtained from 2000 CDC growth charts for the United States. A Standard Deviation Score of 0 represents the population mean. A higher change from baseline in Height SDS indicates a better outcome. The height SDS change from baseline at each visit was modeled using ANCOVA adjusting for baseline age, peak GH levels (log transformed) at diagnosis, delta average-parental height SDS, prior GH dose level (log transformed), and prior GH dose duration (log transformed) as covariates and gender as a factor. Subjects who did not take prior GH treatment were not included in the model.
Time Frame: Baseline and 26 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: standard deviation score
Arm/Group | Lonapegsomatropin
Number analyzed (Participants) | 144
standard deviation score | 0.25 (0.02)

5. Secondary Outcome: Number of Participants With Treatment Emergent Anti-hGH Binding Antibody Formation
Description: Number of participants with treatment emergent anti-hGH antibodies over 26 weeks of weekly lonapegsomatropin (TransCon hGH) treatment. All samples were negative for anti-hGH neutralizing antibodies.
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lonapegsomatropin
Number analyzed (Participants) | 145
Participants | 4

ADVERSE EVENTS:
Time Frame: 26 weeks
Arm/Group | Lonapegsomatropin
All-Cause Mortality (participants affected / at risk) | 0/146
Serious Adverse Events (participants affected / at risk) | 1/146
Other Adverse Events (participants affected / at risk) | 65/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lonapegsomatropin (N=146)
Atrioventricular block (Cardiac disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lonapegsomatropin (N=146)
Pyrexia (General disorders) | 17
Nasopharyngitis (Infections and infestations) | 14
Upper respiratory tract infection (Infections and infestations) | 14
Headache (Nervous system disorders) | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-29): https://cdn.clinicaltrials.gov/large-docs/16/NCT03305016/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT03305016/SAP_001.pdf